CLINICAL TRIAL: NCT01753973
Title: Assessing the Prevalence of Metabolic Syndrome in Renal Transplantation
Status: Completed | Type: Observational
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CAPPesq 164.096
Record Dates: First submitted 2012-12-17; First posted 2012-12-20 (Estimated); Last update posted 2015-12-16 (Estimated); Status verified 2014-06

CONDITIONS: Chronic Renal Failure (CRF); Renal Transplantation
Keywords: Metabolic syndrome; Renal transplantation
MeSH Terms: conditions — Kidney Failure, Chronic; Metabolic Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Metabolic syndrome (MS) is characterized by a series of metabolic and hemodynamic parameters such as hypertension (hypertension), abdominal obesity, dyslipidemia, abnormal glucose metabolism and insulin resistance, resulting in increased cardiovascular morbidity and mortality and the risk for developing type 2 diabetes mellitus (T2DM). Metabolic syndrome is a common event after renal transplantation. The prevalence of MS increases post-transplant with weight gain. In renal transplant recipients, the SM is associated with CVD, diabetes after transplantation, worsening renal function and graft loss. Immunosuppressant medications have primary effect on the pathophysiology of MS. Several studies have evaluated the prevalence and impact of metabolic syndrome in renal transplant recipients as obesity, hypertension, dyslipidemia and use of immunosuppressants. The objectives of this study are to determine whether the determination of the metabolic syndrome at 6 months predicts this same condition at 12 months, determine the prevalence of metabolic syndrome at 12 months, to assess the prevalence of obesity and overweight in this population and to assess the prevalence of diabetes mellitus after renal transplantation. Patients who meet the inclusion criteria and did not meet the exclusion criteria will be invited to participate in the study, signing the Instrument of Consent (IC) and informed about the objectives and procedures of the study to be performed, with age between 18 and 60 years, both sexes, renal transplant recipients Renal Transplant Unit, Hospital das Clinicas, FMUSP living donor or deceased and use of immunosuppressive regimen consisting of tacrolimus, mycophenolate sodium and prednisone. Sampling will be conducted laboratory tests, filling out questionnaires on quality of life and anthropometric measures.

DETAILED DESCRIPTION:
Metabolic syndrome ( MS) is characterized by the presence of a number of metabolic and hemodynamic disorders such as hypertension (HBP ) , abdominal obesity , dyslipidemia, abnormal glucose metabolism and insulin resistance , resulting in increased cardiovascular morbidity and mortality and the risk for developing type 2 diabetes mellitus.

The concept of metabolic syndrome (MS ) was first described by Reaven in 1988 as a combination of obesity , dyslipidemia , hypertension and fasting hyperglycemia , insulin resistance and inflammation as common pathophysiological disorders in cardiovascular disease (CVD). But the first comprehensive definition of MS was established only in 1998 , the World Health Organization ( WHO ) , in order to facilitate research in this area and points as a key indicator of SM the presence of hyperglycemia and / or resistance to insulin associated with days or more metabolic abnormalities (hypertension, dyslipidemia , obesity, and microalbuminuria).

In the general population , the presence of MS is associated with increased risk of developing diabetes mellitus ( DM ) and cardiovascular disease . Some studies have associated the SM to the appearance of proteinuria and reduction in the value of the glomerular filtration rate ( GFR ), suggesting an association SM with chronic kidney disease ( CKD ) .

Metabolic syndrome (MS) consists of complex disorder that involves assembly cardiovascular risk factors related to abdominal fat deposition and insulin resistance . MS is associated with cardiovascular disease , increasing overall mortality by about 1.5 times and cardiovascular mortality by about 2.5 times.

In 2001 , the National Cholesterol Education Program - Panel of the National Cholesterol Education Program ( NCEP - ATP III ), prepared another proposal. According to the NCEP ATP III, SM represents the combination of at least three components.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 60
* Both sexes
* Renal transplant recipients Renal Transplant Unit, Hospital das Clinicas, FMUSP living donor or deceased
* Use of immunosuppressive regimen consisting of tacrolimus, mycophenolate sodium and prednisone

Exclusion Criteria:

* Presence of severe disease with reduced life expectancy
* Presence of diabetic nephropathy
* Presence of cardiac arrhythmia which affects the blood pressure measurement
* Patients with BMI ≥ 40 kg / m²
* Calculated creatinine clearance by Cockroft Gault-≤ 40ml/min
* Transplantation of multiple organs or organ transplant prior to any distinct kidney

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients will be selected by examining the clinical records of Renal Transplant Service, Hospital das Clinicas, Faculty of Medicine, University of São Paulo (HCFMUSP). Patients who meet the inclusion criteria and did not meet the exclusion criteria will be invited to participate in the study, signing the Instrument of Consent (IC) and informed about the objectives and procedures of the study to be performed.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2013-01; Primary Completion 2014-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
To evaluate the prevalence of metabolic syndrome in renal transplant patients. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Elias David-Neto, MD, Principal Investigator — University of Sao Paulo; Fabiana Agena, MS, Principal Investigator — University of Sao Paulo
Locations (1):
- Hospital das Clinicas - Faculdade de Medicina da Universidade de São Paulo, São Paulo, São Paulo, Brazil